CLINICAL TRIAL: NCT06930950
Title: Efficacy of Oral Immunotherapy for Cashew Allergy in Children Aged 1 to 17 Years: a Clinical Prospective Randomized Controlled Interventional Trial
Brief Title: The NACHO Trial (Nut Allergy Children OIT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HUS Skin and Allergy Hospital (Other)
Responsible Party: Principal Investigator, Heidi Sandström, Medical Doctor, HUS Skin and Allergy Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUS/131/2024
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Oral Immunotherapy for Food Allergy; Tree Nut Allergy; Cashew Nut Allergy
Keywords: Oral immunotherapy; Cashew; Tree Nut; Food allergen immunotherapy
MeSH Terms: conditions — Nut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: All patients taking part of the trial will be randomized by simple randomization to the active OIT or control group in a 2:1 manner. Patients will be assigned to a treatment group according to the randomization.
  The control group will crossover to OIT after 12 months of cashew nut avoidance, after a new OFC is done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): The group that will receive oral immunotherapy for cashew nut
  Interventions: Other: Cashew nut oral immunotherapy
- Control group (No Intervention): The group that will continue avoiding cashew nut for 12 months before crossover to active OIT to cashew nut

INTERVENTIONS:
Other: Cashew nut oral immunotherapy — Cashew nut oral immunotherapy (OIT) where the aim is desensitizing individuals with cashew nut allergies. The approach involves the gradual administration of increasing doses of cashew nut protein. The goal of OIT is to increase the threshold of tolerance to cashew nuts, thereby reducing the risk of severe allergic reactions upon accidental exposure
  Arms: Intervention group

SUMMARY:
Most food allergies that begin in early childhood are mild and resolve by school age, but nut allergies persist in about 80-90% of individuals into adulthood. The consumption of nuts, particularly cashew nuts, has increased dramatically in Finland in the 21st century, leading to a rise in severe allergic reactions to cashew nuts among young children. Of the food anaphylaxis cases reported in the Finnish Anaphylaxis Registry between 2015-2020, 49% were caused by nuts, with cashew nuts being the most common trigger. The standard treatment for nut allergies is strict avoidance of nuts and symptom management with emergency medications.

Oral immunotherapy (OIT) is a food allergy treatment that increases tolerance, and it has primarily been studied in school-aged children, with desensitization achieved in about 80% of cases. Permanent tolerance, depending on the allergen, develops in 30-50% of cases within five years. International guidelines recommend peanut OIT for children over the age of 4 who have severe peanut allergies. The likelihood of achieving tolerance, especially permanent tolerance, appears to improve the earlier the treatment is started. To date, only one study (NUIT CRACKER) has been published on cashew nut desensitization in children over 4 years old, involving 50 children, where 88% achieved desensitization to both cashew nuts and pistachios.

The aim of this study is to develop a cashew nut desensitization protocol and investigate its effectiveness in achieving tolerance and permanent desensitization in children aged 1-17 years, compared to cashew nut avoidance. The study will assess the safety of cashew nut desensitization and its impact on the quality of life of patients and their families.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 months - 17 years
2. Sensitization to cashew nut (allergen-specific IgE or positive skin PRICK test)
3. Positive oral food challenge for cashew nut

Exclusion Criteria:

1. Poor adherence
2. Uncontrolled or severe asthma
3. Uncontrolled active or severe or atopic dermatitis
4. Chronic urticaria
5. Eosinophilic esophagitis or other gastrointestinal eosinophilic disorders
6. Active malignant neoplasia
7. Active systemic, autoimmune disease
8. Diabetes treated with insulin
9. Severe systemic illness or severe medical conditions such as cardiovascular or lung diseases
10. Medication with beta blockers
11. Medication with ACE-inhibitors
12. Mastocytosis
13. Pregnancy or breastfeeding
14. Language barriers (not fluent Finnish or Swedish)

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2029-11-05 (Estimated); Study Completion 2029-11-05 (Estimated)

PRIMARY OUTCOMES:
Desensitization | 12 months
  The proportion of patients able to tolerate the target dose of 1000 mg of cashew nut protein in an Oral Food Challenge (OFC) after 12 months of Oral Immunotherapy (OIT) compared to the control group.

SECONDARY OUTCOMES:
Sustained unresponsiveness | 24 months
  The proportion of patients able to tolerate 1000mg of cashew nut protein in an OFC after 23 months of OIT followed by one month of avoidance.
Partial desensitization at 12 months | 12 months
  The proportion of patients able to tolerate a dose below 1000mg of cashew nut protein in an OFC after 12 months of OIT compared to the control group.
Partial desensitization at 24 months | 24 months
  The proportion of patients able to tolerate a dose below 1000 mg of cashew nut protein in an OFC after 23 months of OIT followed by one month of avoidance
Impact on quality of life | 24 months
  The proportion of patients who report improved quality of life in the FAQLQ surveys after OIT, compared to their QoL while avoiding cashew nuts

CONTACTS AND LOCATIONS:
Locations (1):
- HUS Skin and Allergy Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No